CLINICAL TRIAL: NCT03911414
Title: An Open-Label Clinical Trial Conducted Via Telepsychiatry of Complementary and Alternative Treatments (Omega-3 Fatty Acids and Inositol vs. N-acetylcysteine) for the Management of Emotional Dysregulation in Youth
Brief Title: A Clinical Trial Via Telepsychiatry of Treatments for the Management of Emotional Dysregulation in Youth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Director of the Pediatric Bipolar Disorder Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P00846
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Mood Disturbance; Mood Disorders; Natural Supplements; Alternative Treatment
MeSH Terms: conditions — Mood Disorders | interventions — Fatty Acids, Omega-3; Inositol; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omega-3 Fatty Acids + Inositol (Experimental): Subjects will be treated with 1020mg QAM + 1020mg QPM of omega-3 fatty acids and inositol based on weight (subjects under 25kg: 1000mg QD; Subjects weighing 25kg or more: 2000mg QD).
  Interventions: Drug: Open-label Treatment with Omega-3 Fatty Acids + Inositol
- N-acetylcysteine (Experimental): Subjects will be treated with N-acetylcysteine capsules (subjects ages 5-12: 1800mg QD; subjects ages 13-17: 2400mg QD) or effervescent tablets (subjects ages 5-12: 1800mg QD; subjects ages 13-17: 2700mg QD) based on age .
  Interventions: Drug: Open-label Treatment with N-acetylcysteine

INTERVENTIONS:
Drug: Open-label Treatment with Omega-3 Fatty Acids + Inositol — Open-label Treatment with Omega-3 Fatty Acids + Inositol
  Arms: Omega-3 Fatty Acids + Inositol
Drug: Open-label Treatment with N-acetylcysteine — Open-label Treatment with N-acetylcysteine
  Arms: N-acetylcysteine

SUMMARY:
This study consists of a 6-week, open-label, randomized clinical trial study to compare efficacy and tolerability of the natural treatments omega-3 fatty acids, inositol, and N-acetylcysteine (NAC) in the treatment of mood dysregulation in children and adolescents (ages 5-17). Subjects will be randomized to one of two arms: 1) omega-3 fatty acids plus inositol or 2) NAC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 5-17 years of age.
* Current symptoms of emotional dysregulation as indicated by combined T-scores on the Child Behavior Checklist > 180 on the Anxiety/Depression + Aggression + Attention subscales.
* Subjects and their caregivers must be English-speaking, and have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and their caregivers must be willing and able to comply with all study procedures.
* Each subject and his/her parent/guardian must understand the nature of the study. The subject's parent/guardian must sign an informed consent document and the subject must sign an informed assent document.
* Subject must be able to swallow pills.
* Subject must have access to a computer with a camera, speaker, microphone, and internet connection.

Exclusion Criteria:

* Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Serious or unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* History of bleeding diathesis, including those with von Willebrand disease.
* Uncorrected hypothyroidism or hyperthyroidism.
* History of sensitivity to omega-3 fatty acids, inositol or NAC. A non-responder or history of intolerance to omega-3 fatty acid, inositol or NAC after 2 months of treatment at adequate doses as determined by the clinician.
* Severe allergies or multiple adverse drug reactions.
* Unstable or untreated seizure disorder.
* DSM-IV substance use, abuse or dependence.
* Judged clinically to be at serious suicidal risk or C-SSRS score ≥ 4.
* Current diagnosis of schizophrenia.
* Current diagnosis or symptoms of psychosis.
* IQ < 70.
* Pregnant or nursing.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Mean Change in the Parent-Young Mania Rating Scale (P-YMRS) Score | Baseline to 6 Weeks
  The YMRS consists of 11 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe). It is used to assess manic symptoms. Scores from each item are summed to obtain the total YMRS score. The YMRS score ranges from 0-60. A higher score means a higher manic state. Questions are asked about the last week. This scale is generally accepted as the main outcome measure in studies of pediatric bipolar disorder and is linked directly to the core symptoms of mania.

SECONDARY OUTCOMES:
Mean Change in the Parent-completed Children's Depression Inventory (CDI) | Baseline to 6 Weeks
  The CDI consists of 27 items quantifying symptoms such as depressed mood, hedonic capacity, vegetative functions, self-evaluation, and interpersonal behaviors. Each item consists of three statements graded in order of increasing severity from 0 to 2; parents select the one that characterized their child's symptoms best during the past 1 week. The item scores are combined into a total depression score, which ranges from 0 to 54. A higher CDI score means a higher depressive state.
Mean Change in the NIMH Clinical Global Improvement scale (CGI) | Baseline to 6 Weeks
  The CGI is a measure of illness severity adapted for specific disorders. It allows rating of mania, depression and overall bipolar disorder illness, as well as other conditions frequently comorbid with bipolar disorder. The severity score ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The improvement score ranges from 1 (very much improved) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No